CLINICAL TRIAL: NCT01655966
Title: Vitamin D in Addition to Pegylated Interferon and Ribavirin Compared to Pegylated Interferon and Ribavirin Alone in the Treatment of Chronic Hepatitis C Genotype 4.
Brief Title: Vitamin D as an add-on Therapy With Pegylated Interferon and Ribavirin for Chronic Hepatitis c
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany Shehab, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAIL002
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Hepatitis c
Keywords: chronic hepatitis c; hcv; vitamin d
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of care (Active Comparator): Group A: comprises 40 treatment-naive chronic hepatitis c patients who will receive the standard of care treatment: peginterferon Alfa 2a 160 ug once weekly and weight-based ribavirin 1000 or 1200 mg/day (based on body weight < 75 kg or ≥ 75 kg, respectively) in divided doses for 48 weeks.
  Interventions: Drug: pegylated interferon + ribavirin
- Triple therapy (Experimental): Group B: comprises 40 treatment-naive chronic HCV patients who will receive oral vitamin D 1mcg once daily plus peginterferon alfa-2a (160ug once weekly) and weight-based ribavirin 1000-1200 mg daily (based on body weight < 75 kg or ≥ 75 kg, respectively) in divided doses for 48 weeks.
  Interventions: Drug: vitamin D +pegylated interferon + ribavirin

INTERVENTIONS:
Drug: vitamin D +pegylated interferon + ribavirin — Vitamin D: 1mcg once daily 48 weeks Pegylated interferon 160ug once weekly 48 weeks Ribavirin(> 75kg:1200 mg, <75kg:1000mg daily)48 weeks
  Arms: Triple therapy
Drug: pegylated interferon + ribavirin — pegylated interferon 160ug once weekly Ribavirin (> 75kg:1200 mg, <75kg:1000mg daily)48 weeks
  Arms: Standard of care

SUMMARY:
Chronic hepatitis C is endemic in Egypt with a high prevalence of the resistant genotype 4. Conventional standard of care treatment has modest response with only 50% sustained virologic response. Recent reports have suggested an augmented response with the addition of vitamin D. This is a prospective randomized trial to assess the effectiveness of adding vitamin D to standard of care for chronic hepatitis C genotype 4.

ELIGIBILITY:
Inclusion Criteria:

* Adult (male or female), 18 to 65 years of age, with chronic HCV infection
* Liver biopsy showing chronic hepatitis with significant fibrosis using Ishak scoring system
* Compensated liver disease; serum bilirubin < 1.5 mg/dl, INR no more than 1.5, serum albumin > 3.4, platelet count > 75,000 mm, and no evidence of hepatic decompensation (hepatic encephalopathy or ascites)
* Acceptable hematological and biochemical indices (hemoglobin 12.5g/dl for men and 12 g/dl for women; neutrophil count 1500/mm3 or more and serum creatinine < 1.5 mg/dl
* Patients must be serum hepatitis B surface antigen (HBsAg) negative
* Negative Antinuclear Antibodies (ANA) or titer of < 1:160
* Serum positive for anti-HCV antibodies and HCV-RNA
* Abdominal Ultrasound obtained within 3 months prior to entry in the study
* Electrocardiogram for men aged > 40 years and for women aged > 50 years
* Normal fundus examination
* Proper contraception measure throughout the course of treatment and six months later
* Female patients must not breast feed during therapy

Exclusion Criteria:

* Patients who previously received interferon
* HgbA1c > 7.5 or history of diabetes mellitus
* BMI > 34
* Women who are pregnant or breast-feeding
* Males whose female partners are either pregnant or of child-bearing potential or not using birth control and are sexually active
* Other causes of liver disease including autoimmune hepatitis
* Transplant recipients receiving immune suppression therapy
* Screening tests positive for anti-HAV IgM Ab, HBsAg, anti-HBc IgM Ab or anti-HIV Ab
* Decompensated cirrhosis, history of variceal bleeding, ascites, hepatic encephalopathy, CTP score > 6 or MELD score > 8
* Absolute neutrophil count < 1500 cells/mm3; platelet count < 135,000 cells/mm3; hemoglobin < 12 g/dL for women and < 12.5 g/dL for men; or serum creatinine concentration ≥ 1.5 times ULN
* Hypothyroidism or hyperthyroidism not effectively treated with medication
* Alcohol consumption of > 40 grams per day or an alcohol use pattern that will interfere with the study
* History or other clinical evidence of significant or unstable cardiac disease
* History or other clinical evidence of chronic pulmonary disease associated with functional impairment
* Serious or severe bacterial infection(s)
* History of severe or uncontrolled psychiatric disease, including severe depression, history of suicidal ideation, suicidal attempts or psychosis requiring medication and/or hospitalization
* History of uncontrolled severe seizure disorder
* History of immunologically mediated disease requiring more than intermittent anti-inflammatory medications for management or that requires frequent or prolonged use of corticosteroids
* Patients with clinically significant retinal abnormalities

  * Subjects receiving vitamin D for any other medical condition.
  * Subjects with significant active rheumatologic or orthopaedic conditions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-02 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Sustained virologic response | 72 weeks
  Undetectable HCV-RNA 24 weeks after end of treatment.

SECONDARY OUTCOMES:
rapid virologic response | 4 weeks
  undetectable HCV-RNA 4 weeks after commencement of treatment
End-of-treatment response | 48 weeks
  undetectable HCV-RNA 48 weeks after commencement of treatment
Adverse events | 72 weeks
  Adverse events that could be reasonably and temporally associated with administration of drugs
early virologic response | 12 weeks
  Early virologic response: undetectable HCV-RNA 12 weeks after commencement of treatment.
  Partial early virologic response: decrease of more than 2login HCV-RNA.
  No early virologic response: increase, stationary or decreased less than 2log HCV-RNA.

CONTACTS AND LOCATIONS:
Overall Officials: Tamer Elbaz, MD, Principal Investigator — Cairo University; Hany Shehab, MD, Study Director — Cairo University
Locations (1):
- National Railway Hospital Center, Cairo, Egypt